CLINICAL TRIAL: NCT05479123
Title: Assessing the Impact of Dosage Frequency of Propranolol on Sleep Patterns in Patients With Infantile Hemangiomas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Matthew Greives, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-22-0246
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Infantile Hemangioma
MeSH Terms: conditions — Hemangioma, Capillary | interventions — Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ter in die (TID)three times a day (Experimental)
  Interventions: Drug: Propranolol three times a day
- bis in die (BID)twice a day (Experimental)
  Interventions: Drug: Propranolol twice a day
- Control (Active Comparator)
  Interventions: Drug: Timolol

INTERVENTIONS:
Drug: Propranolol three times a day — Patients with larger (>2cm) or multiple (>1) hemangiomas in this arm will get propranolol in the following regimen:
  Week 1: 0.5 mg/kg/day divided TID Week 2: 1 mg/kg/day divided TID Week 3: 2 mg/kg/day divided TID. Patients will stay on this dosage until their 3 month follow up visit.
  Arms: ter in die (TID)three times a day
Drug: Propranolol twice a day — Patients with larger (>2cm) or multiple (>1) hemangiomas in this arm will get propranolol in the following regimen:
  Week 1: 0.5 mg/kg/day divided BID Week 2: 1 mg/kg/day divided BID Week 3: 2 mg/kg/day divided BID. Patients will stay on this dosage until their 3 month follow up visit.
  Arms: bis in die (BID)twice a day
Drug: Timolol — Patients with a small (<2cm) isolated infantile hemangioma are prescribed timolol 0.5% ophthalmic drops, a topical beta-blocker(1 drop BID directly onto the hemangioma).
  Arms: Control

SUMMARY:
The purpose of this study is to assess the baseline sleep pattern disruption for patients starting oral propranolol at the standard BID dosing regimen compared to the control (timolol) group and to determine if there is a significant improvement in the sleep patterns in infants taking oral propranolol on the TID dosing regimen versus the control (timolol) group

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed hemangiomas.
* English or Spanish speaking only

Exclusion Criteria:

* Parents who do not consent to the study.
* Significant cardiac or pulmonary disease who are unable to tolerate oral propranolol

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of sleep awakenings per night as assessed by the Brief Infant Sleep Questionnaire(BISQ) | 6 months from baseline

SECONDARY OUTCOMES:
Total amount of time subject is awake at night | 3 months from baseline
Total amount of time subject is awake at night | 6 months from baseline
Total amount of time subject is awake at night | 9 months from baseline
Total amount of time subject is awake at night | 12 months from baseline
Total amount of time subject is awake at night | 15 months from baseline
Total amount of time subject is awake at night | 18 months from baseline
Qualitative assessment of difficulty falling asleep as assessed by the Brief Infant Sleep Questionnaire(BISQ) | 3 months from baseline
  will be assessed categorically from very easy, somewhat easy, neither easy nor difficulty, somewhat difficult or very difficult.
Qualitative assessment of difficulty falling asleep as assessed by the Brief Infant Sleep Questionnaire(BISQ) | 6 months from baseline
  will be assessed categorically from very easy, somewhat easy, neither easy nor difficulty, somewhat difficult or very difficult.
Qualitative assessment of difficulty falling asleep as assessed by the Brief Infant Sleep Questionnaire(BISQ) | 9 months from baseline
  will be assessed categorically from very easy, somewhat easy, neither easy nor difficulty, somewhat difficult or very difficult.
Qualitative assessment of difficulty falling asleep as assessed by the Brief Infant Sleep Questionnaire(BISQ) | 12 months from baseline
  will be assessed categorically from very easy, somewhat easy, neither easy nor difficulty, somewhat difficult or very difficult.
Qualitative assessment of difficulty falling asleep as assessed by the Brief Infant Sleep Questionnaire(BISQ) | 15 months from baseline
  will be assessed categorically from very easy, somewhat easy, neither easy nor difficulty, somewhat difficult or very difficult.
Qualitative assessment of difficulty falling asleep as assessed by the Brief Infant Sleep Questionnaire(BISQ) | 18 months from baseline
  will be assessed categorically from very easy, somewhat easy, neither easy nor difficulty, somewhat difficult or very difficult.
Amount of time it takes for subject to fall asleep | 3 months from baseline
Amount of time it takes for subject to fall asleep | 6 months from baseline
Amount of time it takes for subject to fall asleep | 9 months from baseline
Amount of time it takes for subject to fall asleep | 12 months from baseline
Amount of time it takes for subject to fall asleep | 15 months from baseline
Amount of time it takes for subject to fall asleep | 18 months from baseline
Longest stretch of time the subject is asleep without waking up | 3 months from baseline
Longest stretch of time the subject is asleep without waking up | 6 months from baseline
Longest stretch of time the subject is asleep without waking up | 9 months from baseline
Longest stretch of time the subject is asleep without waking up | 12 months from baseline
Longest stretch of time the subject is asleep without waking up | 15 months from baseline
Longest stretch of time the subject is asleep without waking up | 18 months from baseline
Clinical Response to Medication as assessed by the qualitative clinical assessment on size, color changes of hemangiomas | 3 months from baseline
Clinical Response to Medication as assessed by the qualitative clinical assessment on size, color changes of hemangiomas | 6 months from baseline
Clinical Response to Medication as assessed by the qualitative clinical assessment on size, color changes of hemangiomas | 9 months from baseline
Clinical Response to Medication as assessed by the qualitative clinical assessment on size, color changes of hemangiomas | 12 months from baseline
Clinical Response to Medication as assessed by the qualitative clinical assessment on size, color changes of hemangiomas | 15 months from baseline
Clinical Response to Medication as assessed by the qualitative clinical assessment on size, color changes of hemangiomas | 18 months from baseline
Number of participants with side effects | 18 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Greives, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No